CLINICAL TRIAL: NCT01008332
Title: An Escalating, Multiple-dose Study in House Dust Mite Allergic Subjects to Assess the Safety of Intradermal Injection of ToleroMune HDM
Brief Title: Safety of ToleroMune House Dust Mite (HDM) to Treat House Dust Mite Allergy in HDM Allergic Subjects With Rhinoconjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Circassia Limited (Industry)
Collaborators: Adiga Life Sciences, Inc. (Industry)
Responsible Party: Dr Rod Hafner, VP R&D, Circassia Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TH001
Record Dates: First submitted 2009-11-04; First posted 2009-11-05 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2010-11

CONDITIONS: Allergy
Keywords: House Dust Mite Allergy; Immunotherapy; Rhinoconjunctivitis; Toleromune HDM
MeSH Terms: conditions — Hypersensitivity; Dust Mite Allergy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental): ToleroMune HDM, subjects to receive either active or placebo comparator
  Interventions: Biological: Toleromune HDM; Biological: Placebo
- Cohort 2 (Experimental): ToleroMune HDM, subjects to receive either active or placebo comparator
  Interventions: Biological: Toleromune HDM; Biological: Placebo
- Cohort 3 (Experimental): ToleroMune HDM, subjects to receive either active or placebo comparator
  Interventions: Biological: Toleromune HDM; Biological: Placebo
- Cohort 4 (Experimental): ToleroMune HDM, subjects to receive either active or placebo comparator
  Interventions: Biological: Toleromune HDM; Biological: Placebo
- Cohort 5 (Experimental): Toleromune HDM, subjects to receive either active or placebo comparator
  Interventions: Biological: Toleromune HDM; Biological: Placebo

INTERVENTIONS:
Biological: Toleromune HDM — ToleroMune HDM dose 1x4 administrations 4 weeks apart
Biological: Placebo — Placebo comparator, 1x4 administrations 4 weeks apart

SUMMARY:
The prevalence of allergic sensitisation to House Dust Mite (HDM) varies from region to region and depends on the regional prevalence of HDM. In the third National Health and Nutrition Examination Surveys, 54.3% of the US population had positive test responses to one or more allergens, with the prevalence for HDM being 27.5%. Like many other allergens, exposure to HDMA in sensitised patients is associated with poorer lung function, greater medication requirements and more asthma symptoms as well as chronic rhinosinusitis symptoms.

ToleroMune HDM is a novel, synthetic, allergen-derived peptide desensitising vaccine, currently being developed for the treatment of Houst Dust Mite allergy.

The purpose of the present study is to evaluate the safety and tolerability of multiple ascending doses of ToleroMune HDM in subjects in subjects with a documented history of allergic rhinoconjunctivitis on exposure to house dust mite. The efficacy of ToleroMune HDM will also be explored in these subjects using the Late Phase Skin Response, Early Phase Skin Response and Conjunctival Provocation Test.

DETAILED DESCRIPTION:
This study is designed as a randomised, double-blind, placebo-controlled study to evaluate the safety and tolerability of escalating multiple doses of ToleroMune HDM in subjects with a documented history of allergic rhinoconjunctivitis on exposure to house dust mite. The efficacy of ToleroMune HDM will also be explored in these subjects using the LPSR, EPSR, CPT and levels of HDM specific IgE. A single centre will be initiated first, with a second centre included as a backup, if needed, to enable recruitment numbers to be met.

The study will consist of 3 study periods. In Period 1, Screening will be performed up to a maximum of 8 weeks before randomisation and may consist of one or two visits to the clinic, at the Investigator's discretion. Baseline Challenge will consist of a single visit 1 to 4 weeks before randomisation.

Period 2 (Treatment Period) will consist of 4 visits (Visits 3A-3D) four weeks apart (28±2 days). Subjects who comply with the inclusion/exclusion criteria will be assigned to one of 5 dose groups. The first dose group will receive 4 administrations of ToleroMune HDM. Successive dose groups will increasing doses given as 4 administrations of ToleroMune HDM, provided the first administration of the previous dose was safe and well tolerated.

In Period 3, Post-treatment Challenge will take place 18-22 weeks after the first administration in the Treatment Period. Assessments performed will be identical to those at the Baseline Challenge. Follow-up will be conducted 3-10 days after PTC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-65 years
* Miniumum 1 year history of rhinoconjunctivitis on exposure to HDM
* Positive skin prick test to whole Der p allergen
* LPSR to whole Der p allergen 8-10 hours after intradermal injection of greater than 35mm diameter response
* Positive CPT to whole Der p allergen with a score ≥4

Exclusion Criteria:

* Subjects with a history of asthma
* Subjects with an FEV1 <80% of predicted
* Subjects with a Der f or Der p specific IgE >100 kU/L
* Subjects with an acute phase skin response to whole Der p or whole Der f allergen with a mean wheal diameter > 50 mm
* Subjects who score >1 for redness of conjunctiva or who have any watering or itchiness in the eye before administration of the CPT
* Treatment with beta-blockers, alpha-adrenoreceptor blockers, tranquillizers or psychoactive drugs
* History of any significant disease or disorder (e.g. cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, malignant, psychiatric, major physical impairment)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of multiple intradermal injections of ToleroMune HDM in HDM allergic subjects with allergic rhinoconjunctivitis | 18-22 weeks

SECONDARY OUTCOMES:
Mean change from baseline in area of the LPSR 8 hours after intradermal challenge with whole HDM allergen at PTC after ToleroMune HDM injection compared to placebo | 18-22 weeks
Mean change from baseline in area of the EPSR 15 minutes after intradermal challenge with whole HDM allergen at PTC after ToleroMune HDM injection compared to placebo | 18-22 weeks
Mean change from baseline in CPT score at PTC after ToleroMune HDM injection compared to placebo | 18-22 weeks
Mean change from baseline in concentration of HDM specific IgE at PTC after ToleroMune HDM injection compared to placebo | 18-22 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Hebert, MD, Principal Investigator — Centre de Recherche Appliqué en Allergie de Québec
Locations (1):
- Centre de Recherche Appliqué en Allergie de Québec, Québec, Quebec, Canada